CLINICAL TRIAL: NCT04723264
Title: The Development of Eating Behavior in Infancy: Associations With Behavior, Diet, and Growth at School Age
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Julie Lumeng, Thomas P Borders Family Research Professor of Child Behavior and Development, Professor of Pediatrics, Associate Dean for Research, Medical School, Professor of Nutritional Sciences, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00181248; R01HD084163 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Eating Behavior
Keywords: Body mass index; Dietary quality; Children
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eating behavior activities (Experimental)
  Interventions: Behavioral: Food protocols

INTERVENTIONS:
Behavioral: Food protocols — Participants will engage in several activities (i.e. offering a variety of foods and age appropriate games, etc.) regarding eating behaviors.
  Participants will be asked to videotape interactions using a secure system. An alternative option may be provided if this videotaping is not acceptable.

SUMMARY:
This study will examine children's eating behavior. The study will enroll approximately 400 participants (200 child/parent pairs).

At certain time points, participants will engage in activities involving the presentation of food and the observation of behavioral responses to these presentations, as well as the completion of questionnaires

DETAILED DESCRIPTION:
This research study is a complex, long term investigation of the relationships between children's eating behaviors, and parent-child interaction during eating and their associations with BMI and dietary intake. It builds on earlier observational research which, like this research, had small experimental components used to classify children into different phenotypic groups based on different responses to the experimental conditions. The small activities and experiments of this follow up study constitute a trial as defined by NIH, registered here. The exploratory outcomes measured from these activities are not listed in this registration for reasons of scientific integrity. To be clear, the bigger structure of this research is essentially an observational follow up study with the same children who were previously studied as infants. The goal of the project is to identify potential future intervention targets.

ELIGIBILITY:
Inclusion Criteria for Children (ages 5-7.99) and their parents (18 and older):

* Prior participation in "The Development of Eating Behavior in Infancy" project
* Family lives within reasonable driving distance of the University of Michigan

Exclusion Criteria:

* Significant developmental delays that would impede child's ability to participate
* Foster child
* Child has developed significant health problems that affect appetite, eating, or growth.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index z - score (BMIz) | 1- 2 years
  Children will be weighed and measured using a portable stadiometer. BMI will be calculated and child BMI z-score derived using age- and sex-specific norms from Centers for Disease Control and Prevention (CDC) growth charts.

SECONDARY OUTCOMES:
Dietary Intake | 1- 2 years
  Mean dietary intake of macro- and micro-nutrients using an automated self-administered 24-hour dietary assessment tool across two recall days.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lumeng, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The research will generate demographic, behavioral, videorecorded, and anthropometric data. (Note the researchers will not make video data available). Meta data will also be included in the selected repositories. Of note, this will include only child age, but not birthdate or date of study visit as these would violate confidentiality. The metadata will include the data dictionaries, which describe the generation of all variables.
Supporting Information: Study Protocol, ICF
Time Frame: We will make the de-identified data available within one year of completion of the study at the University of Michigan's data repository (Deep Blue Data Repository). We will not place video/audio data in the data repository due to the inability to de-identify the participants and protect their privacy
Access Criteria: All data in the Deep Blue Data repository are available to anyone for download without restriction.

REFERENCES:
- [Derived] Ventura AK, Ross KJ, Miller AL, DeJesus JM, Tan CC, Lumeng JC. Co-Development of Infant Satiation Cues and Maternal Feeding Behaviors during Infancy. Curr Dev Nutr. 2025 Sep 3;9(10):107542. doi: 10.1016/j.cdnut.2025.107542. eCollection 2025 Oct. PMID 41081012

DOCUMENTS (1):
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT04723264/ICF_000.pdf